CLINICAL TRIAL: NCT03153631
Title: Evaluating Female Sexual Dysfunction in Breast Cancer Patients After Mastectomy
Brief Title: Female Sexual Dysfunction in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanaa H Bery, princilal investigator, Assiut University
Other Study IDs: fsdbc
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Female Breast Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most frequently diagnosed cancer and the leading cause of cancer death among females world wide. breast cancer alone accounts for 25% of all cancer cases and 15% of all cancer deaths among females.

DETAILED DESCRIPTION:
In Egypt, cancer breast is one of the commonest cancers among females representing 38.8%.cancer breast among females ranked the top with a high frequency in lower, middle, upper Egypt (33.8%,26.8%,38.7% resp.).

Women who developed breast cancer were more amenable than women who remained free of breast carcinoma to experience reduced physical function, vitality, social function.

Difficulties related to sexuality and sexual functioning were common and occurred soon after surgical and adjuvant treatment. addressing these problems is essential to improve the quality of life of young women with breast cancer.

Sexuality is a basic and important domain of human experience that can be damaged during and following cancer treatment. The risk of sexual dysfunction is even of greater importance among young cancer patients and survivors, with young breast cancer patients at particularly high risk.

In cancer breast patients, various factors can induce sexual dysfunction. Some of these factors; hormonal alterations induced by chemotherapy and radiotherapy, or physiological and functional disturbances are related to the deterioration of physical condition. These factors are strictly clinical.

Other factors which induce disturbances in sexual behavior, such as anxious\ depressive reactions in adapting to illness and treatment and cancerophobic reactions and loss of self esteem that accompany any illness are more psychological\ psychiatric in nature.

Having sexual problems (or dysfunction) includes experiencing disturbances in sexual desire and physiological changes associated with loss of sexual desire and arousal, reduction in sexual pleasure, difficulty achieving orgasm, anxiety about sexual performance and pain during intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years old.
* Social status: Married.
* (Performance status): Who 0-1

  * 0-Asymptomatic (fully active, able to carry on all predisease activities without restriction)
  * 1-Symptomatic but completely ambulatory (restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature. For example, light housework, office work)

Exclusion Criteria:

* Pregnant women.
* Comorbidities (Diabetes mellitus., Hypertension).
* Female genital tract disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Seventy five female, with cancer breast who did mastectomy at child bearing period, will be recruited from the outpatient clinic of clinical oncology department in Assiut University hospital and South Egypt Cancer Institute.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
assessment of female sexual dysfunction in breast cancer patients after mastectomy using questionaire | one month
  description of manner of female sexual dysfunction after mastectomy using Arabic Female Sexual Function Index and FEMALE SEXUAL FUNCTION INDEX DOMAIN SCORES AND FULL SCALE SCORE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bober SL, Varela VS. Sexuality in adult cancer survivors: challenges and intervention. J Clin Oncol. 2012 Oct 20;30(30):3712-9. doi: 10.1200/JCO.2012.41.7915. Epub 2012 Sep 24. PMID 23008322
- [Background] Chapman RM. Effect of cytotoxic therapy on sexuality and gonadal function. Semin Oncol. 1982 Mar;9(1):84-94. PMID 6176028
- [Background] Derogatis LR, Morrow GR, Fetting J, Penman D, Piasetsky S, Schmale AM, Henrichs M, Carnicke CL Jr. The prevalence of psychiatric disorders among cancer patients. JAMA. 1983 Feb 11;249(6):751-7. doi: 10.1001/jama.249.6.751. PMID 6823028
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Katz RC, Jardine D. The relationship between worry, sexual aversion, and low sexual desire. J Sex Marital Ther. 1999 Oct-Dec;25(4):293-6. doi: 10.1080/00926239908404006. PMID 10546167
- [Background] Fobair P, Stewart SL, Chang S, D'Onofrio C, Banks PJ, Bloom JR. Body image and sexual problems in young women with breast cancer. Psychooncology. 2006 Jul;15(7):579-94. doi: 10.1002/pon.991. PMID 16287197
- [Background] Sadovsky R, Basson R, Krychman M, Morales AM, Schover L, Wang R, Incrocci L. Cancer and sexual problems. J Sex Med. 2010 Jan;7(1 Pt 2):349-73. doi: 10.1111/j.1743-6109.2009.01620.x. PMID 20092444